CLINICAL TRIAL: NCT01003314
Title: A Phase I/IIa Study to Assess the Safety and Immunogenicity of New Malaria Vaccine Candidates AdCh63 MSP1 Alone and With MVA MSP1
Brief Title: A Study of the Safety and Effectiveness of Two New Malaria Vaccines
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Heather House, University of Oxford
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC037
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Malaria
Keywords: Vaccine; Safety; Immunogenicity; Protection; Sporozoite challenge
MeSH Terms: conditions — Malaria | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental)
  Interventions: Biological: AdCh63-MSP1 (lower dose) vaccine and MVA-MSP1 vaccine
- Group 2 (Experimental)
  Interventions: Biological: AdCh63-MSP1 vaccine (higher dose) and MVA-MSP1 vaccine followed by challenge

INTERVENTIONS:
Biological: AdCh63-MSP1 (lower dose) vaccine and MVA-MSP1 vaccine — Group 1A: single dose of AdCh63-MSP1 vaccine 5 x 10^9 vp administered IM. Group 1B: single dose of AdCh63-MSP1 vaccine 5 x 10^9 vp administered IM followed by a single dose of MVA-MSP1 vaccine 5 x 10^8 vp administered IM 8 weeks later
  Arms: Group 1
Biological: AdCh63-MSP1 vaccine (higher dose) and MVA-MSP1 vaccine followed by challenge — Group 2A: single dose of AdCh63-MSP1 vaccine 5 x 10^10 vp administered IM. Group 2B: single dose of AdCh63-MSP1 vaccine 5 x 10^10 vp administered IM followed by a single dose of MVA-MSP1 vaccine 5 x 10^8 vp administered IM 8 weeks later. Group 2C: single dose of AdCh63-MSP1 vaccine 5 x 10^10 vp administered IM followed by a single dose of MVA-MSP1 vaccine 5 x 10^8 vp administered IM 8 weeks later and subsequent sporozoite malaria challenge 12-28 days post second vaccination
  Arms: Group 2

SUMMARY:
This study aims to test the safety of two new malaria vaccines AdCh63 MSP1 and MVA MSP1. These vaccines consist of inactivated viruses which have been modified - so they cannot reproduce (replicate) in humans, and also to include genetic material (genes) for malaria proteins which are expressed by the malaria parasite during blood stage infection. The vaccines are designed to stimulate an immune response to these malaria proteins (immunogenicity describes the nature and magnitude of this immune response), to provide protection against malaria infection. This protection has been demonstrated in nonhuman studies. Although these vaccines have not been given to humans before, similar vaccines using the same viruses with different malaria genes have been given to humans before. In these studies, the vaccines have been shown to be safe. They have also provided evidence from laboratory tests of immunogenicity. In this study the investigators main aim is to ensure these new vaccines given alone and in combination are safe. The investigators will increase the dose of the first vaccine (AdCh63 MSP1) given to volunteers if the initial dose is safe. The investigators also wish to ensure that challenging a small number of volunteers who have received both vaccines with malaria infection from the bites of infected mosquitos(sporozoite challenge) is safe. Sporozoite challenge has been widely used in humans to test the effectiveness of malaria vaccines and is considered a well established, reliable, predictable and safe system.In the study the investigators will also look for evidence of immunogenicity of these new vaccines, and whether there is any delay to developing malaria following sporozoite challenge. The study will be conducted at the University of Oxfords Centre for Clinical Vaccinology and Tropical Medicine (CCVTM). The challenge part of the study will take place at the insectary at Imperial College, (Infection and Immunity Section)in London.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* For females only, willingness to practice continuous effective contraception during the study and a negative pregnancy test on the day(s) of vaccination and/or challenge
* For males only, willingness to use barrier contraception until 3 months after last vaccination
* Agreement to refrain from blood donation during the course of the study
* Written informed consent

Exclusion Criteria:

Significant concern raised by GP in relation to participation

* Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of a recombinant adenoviral and/or MVA-vectored vaccine
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days)immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products, Kathon
* History of clinically significant contact dermatitis
* A predicted ten year risk of fatal cardiovascular disease of =>5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system [59]
* History of arrhythmia or congenital QT interval prolongation
* Family history of sudden cardiac death
* Contraindication to both anti-malarial drugs (Riamet and chloroquine)

  o concomitant use with other drugs known to cause QT-interval prolongation, (e.g. macrolides, quinolones, amiodarone etc)
* Any history of anaphylaxis in reaction to vaccination
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Any other significant disease, disorder or finding, which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or may influence the result of the study, or the volunteer's ability to participate in the study
* Any history of malaria
* Travel to a malaria endemic region during the study period or within the previous six months
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
* Any other finding which in the opinion of the investigators would significantly increase the risk of having an adverse outcome from participating in the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety of new candidate malaria vaccines AdCh63 MSP1 administered alone, and with MVA MSP1 in a prime-boost regime, to healthy volunteers. and safety of the prime-boost vaccine strategy following malaria sporozoite challenge. | Up to 6 months post enrollment into the study

SECONDARY OUTCOMES:
Humoral and cellular immune responses generated by AdCh63 MSP1, when administered to healthy volunteers alone, with MVA MSP1, and following sporozoite challenge. Efficacy of AdCh63 MSP1 and MVA MSP1 against malaria sporozoite challenge | Up to 6 months post enrollment into the study

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, D.Phil, FRCP, Principal Investigator — Univeristy of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, University of Oxford, Oxford, United Kingdom